CLINICAL TRIAL: NCT05693311
Title: Inflammatory Bowel Disease Related Joint Manifestations Including the Incidence, Types, Relation to Disease Activity and Types of Treatment
Brief Title: Inflammatory Bowel Disease Related Joint Manifestations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Youstina Yosry Soliman (Other)
Responsible Party: Sponsor-Investigator, Youstina Yosry Soliman, resident doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Joint manifestations in IBD
Record Dates: First submitted 2022-12-24; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: IBD; Joint Diseases
Keywords: IBD; periphral and axial spondylopathy
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this research is to identify incidence of jiunt manifestations by its both types axial and periphral in IBD patients, its types , relation to IBD activity, lines of treatment using and how they are effective in prevention and in treatment of these joint manifestations.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic immune-mediated disorder divided into two large types Crohn disease and ulcerative colitis. Crohn disease may affect any part of the gastrointestinal tract (GIT), whereas Ulcerative colitis affects the large intestine . IBD is also described to cause remissions and relapses or activity. IBD is a multisystem condition that affects mainly the gastrointestinal, musculoskeletal, ocular, and cutaneous systems. Those complications that arise outside the intestinal inflammation are known as extra intestinal manifestations (EIMs) of IBD, EIMs present in 5% to 50% of all IBD patients these may be :skin, eyes, kidneys, liver, anaemia.

In a focused point musculoskeletal manifestations being the most common EIM with a incidence about 40%. It was divided into:

A. Axial type (spondyloarthropathy) B. Peripheral type divided into : 1.Type 1 (pauciarticular). 2.Type 2 (polyarticular) In this research we shall focus on the confirmed data for diagnosis of IBD by history , lab investigations & colonoscopy and biopsy including disease location . Then onset of joint manifestations in relation to both intestinal & other extra intestinal manifestations . The effect of disease activity on routine lab investigations including CBC, kidney function , liver function , ESR, CRP & on imaging like x-ray .

Also the effect of disease activity on joint manifestations is an important point to be discussed .

For this purpose, a validated detailed questionnaire according to farisoğullari 2021 consisting of six questions was asked (1). Have you ever had swelling or pain in fingers , toes or any other joint with no apparent reason? (2).Has an entire finger or toe becomes swollen, making it look like a 'sausage' ? (3). Have you had pain in your heels? (4). Have you ever had back pain lasting at least 3 months that was not injury related? (5). Do you have low back pain in the morning after resting that improves with exercise? (6). Do you wake up at night because of low back pain?.

The response of joint manifestations to different routes of treatment of IBD is also of great importance , A good response of back pain to a full dose of non-steroidal anti-inflammatory drugs was defined as "not anymore present "or "much better". Immunomodulators have been efficacious in patients with peripheral arthritis and other extra-intestinal manifestations, but they are not effective for the treatment of axial symptoms of spondylitis.

The treatment of peripheral involvement and/or enthesitis and/or dactylitis is based on local steroid injections, while sulfasalazine and/or low doses of systemic steroids may be useful in case of inadequate response to intra-articular steroids. Sulfasalazine induces only a little improvement in peripheral arthritis. Immunomodulators such as methotrexate, azathioprine, cyclosporine and leflunomide were also effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed by colonoscopy and biopsy of IBD either crhons disease or ulcerative colitis from2017 to 2022 attending IBD clinic in EL-RAGHY LIVERHOSPITAL.

Exclusion Criteria:

* Patients with a known diagnosis of any other joint disease like:

  1. autoimmune disease like SLE , RA , psoriasis
  2. Osteoarthritis
  3. Gouty arthritis
  4. Malignancy
  5. Polymyalgia rheumatica

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with inflammatory bowel disease attending IBD clinic in EL-RAGHY LIVERHOSPITAL.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The joint manifestations in Inflammatory bowel disease patients. | 2017 to 2024
  The main purpose of this research is to identify incidence of joint manifestations by its both types axial and peripheral in crohns disease and ulcerative colitis patients, relation to the disease activity,other extra intestinal manifestations, lines of treatment used and how they are effective in prevention and in treatment of these joint manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ali, ass.prof doc, Study Director — assiut univeristy

REFERENCES:
- [Background] Voulgari PV. Rheumatological manifestations in inflammatory bowel disease. Ann Gastroenterol. 2011;24(3):173-180. PMID 24713717
- [Background] Fragoulis GE, Liava C, Daoussis D, Akriviadis E, Garyfallos A, Dimitroulas T. Inflammatory bowel diseases and spondyloarthropathies: From pathogenesis to treatment. World J Gastroenterol. 2019 May 14;25(18):2162-2176. doi: 10.3748/wjg.v25.i18.2162. PMID 31143068
- [Background] Di Carlo M, Luchetti MM, Benfaremo D, Di Donato E, Mosca P, Maltoni S, Benedetti A, Gabrielli A, Grassi W, Salaffi F. The DETection of Arthritis in Inflammatory boweL diseases (DETAIL) questionnaire: development and preliminary testing of a new tool to screen patients with inflammatory bowel disease for the presence of spondyloarthritis. Clin Rheumatol. 2018 Apr;37(4):1037-1044. doi: 10.1007/s10067-017-3937-6. Epub 2017 Dec 4. PMID 29204760